CLINICAL TRIAL: NCT03873896
Title: The Skin Wrinkle Test: a Simple Clinical Test of Regional Block Success
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Peter Collins, Peter Collins, Assistant Professor, Principal Investigator, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 20190762
Record Dates: First submitted 2018-09-06; First posted 2019-03-14 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Skin Manifestations
MeSH Terms: conditions — Skin Manifestations

STUDY DESIGN:
Intervention Model Description: Blinded control trial assessing aquagenic skin wrinkling after digital nerve blockade in healthy volunteers. Digital nerve blocks to be performed on the left or right ring fingers of volunteers (to be randomized with coin toss) with the unblocked finger of each volunteer acting as its own control
Who Masked: Outcomes Assessor
Masking Description: Photos of blocked digits will be taken and presented to blinded assessors to rate on a pre-determined scale of wrinkling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blocked finger (Experimental): The experimental arm will be the ring finger of the volunteer that is blocked (randomized either right or left hand) with a digital nerve block (described elsewhere in the submission). The skin wrinkle test (diagnostic test) will be applied to this arm
  Interventions: Diagnostic Test: Stimulated skin wrinkling test; Procedure: Digital Nerve Block
- Unblocked finger (Active Comparator): The control arm will be the finger of the same volunteer that is not under the influence of digital nerve block. This will be the corresponding digit (the ring finger) on the opposite hand of the side that was blocked (determined by coin toss). The skin wrinkle test (diagnostic test) will be applied to this arm
  Interventions: Diagnostic Test: Stimulated skin wrinkling test

INTERVENTIONS:
Diagnostic Test: Stimulated skin wrinkling test — Stimulated skin wrinkling induced by the application of EMLA (eutectic mixture of local anesthetic) cream to the finger pads of blocked and unblocked fingers of study volunteers (test applied to both study arms)
Procedure: Digital Nerve Block — A digital nerve block is performed by injecting a total of 3 millilitres of 2% Lidocaine at the base of the ring finger of randomized hand of the volunteer. The effect of the block is confirmed clinically before proceeding with the study data collection. Please see the description for more details on the procedure
  Arms: Blocked finger

SUMMARY:
Wrinkling of the hands and feet with exposure to moist environments is a commonly observed phenomenon. This "stimulated skin wrinkling" (SSW) is the result of direct stimulation of digital nerve sympathetic fibers. The resulting effect is a sympathetically mediated vasoconstriction with loss of finger pulp volume, overlying skin traction and wrinkling. It has been established that multiple disease states of the sympathetic nervous system such as diabetic neuropathy, leprosy and nerve injury can lead to impaired SSW of the affected limb. While this test has been successfully utilized for over 80 years to assess patients with sympathetic pathology, it has never been evaluated as a tool to determine the success of a regional nerve block. A regional nerve block is a method of anesthesia that involves injecting a local anesthetic around a particular nerve or nerve bundle in order to block the sensation of pain from that particular body part.

This is of particular importance in the paediatric or non verbal population. These patients may not be able to reliably confirm the effectiveness of their analgesia. Pediatric anesthesiologists often perform these regional blocks on already anesthetized children whereas the non-verbal or cognitively impaired population may not be able to verbalize block effectiveness.

This test, if proven effective as a means of determining block success, would be a quick, non-invasive and inexpensive method of ensuring adequate intra-operative and post operative analgesia for patients. As this is a pilot project focused on establishing the SSW test as an effective tool for assessing regional block success on awake volunteers, further studies would need to be performed to assess test effectiveness in different clinical situations.

DETAILED DESCRIPTION:
We estimated the sample size of four based on the use of a non-parametric analysis, and for the purpose to keep the sample of subjects to a minimum. Further that the effect size is expected to be a large effect (e.g. as it's a binary response yes/no wrinkling, previous experience and literature with the use of the cream for obtaining a pronounced effect of wrinkling (4-5) on the PING scale for an individual with normal peripheral nerve response on an unblocked digit. By using the non-parametric chi square statistical analysis it does not rely on means and standard deviation so it is more sensitive to even small differences beyond chance.

After informed written consent is obtained, volunteers will be subjected to a digital nerve block of ring finger of either the left or right hands. The hand to be blocked will be randomized using a coin toss. The nerve block will be performed by members of the research team with extensive experience in regional blockade. After full sterile preparation, 3 cc's of 2% plain lidocaine will be used to perform the digital nerve block. Five minutes after the performance of the block, the affected digit will be tested by both light touch and temperature to confirm block success. Ring fingers of both hands of the volunteer will then be wrapped in an occlusive dressing after 1mL (millilitre) of EMLA (Eutectic Mixture of Local Anesthetic) cream is applied to the pad of each finger. Photos of the blocked finger as well as the corresponding unblocked finger of the opposite hand will be taken with tangential lighting at 0, 10, 20 and 30 minutes from the time of exposure to EMLA cream. The EMLA cream and occlusive dressings will be removed for each photo then reapplied after the photo is completed. Photos will then be evaluated by two members of the research team blinded as to the finger blocked in each volunteer. Evaluators reviewing the photos of individual fingers will be asked to grade the degree of wrinkling on a scale from 0 to 4 described by Ping Ng et al (a previously established scale to assess stimulated skin wrinkling).

Clinical Care Measures To ensure safety of the study participants, digital nerve blocks will be performed by anesthesiologists or anesthesiology residents with experience in performing these blocks and under strict aseptic conditions. A limited amount of lidocaine is utilized to ensure adequate block but minimize duration of block as well as risks of toxicity. The study participants will be fully monitored with continuous 3 lead ECG, NIBP (non-invasive blood pressure) measurements every 5 minutes and continuous pulse oximetry for 120 minutes period after the analysis. The participants will be attended by at least one physician for this entire period. A follow up telephone call will be performed 24 hours after the performance of the digital nerve block to assess for complications.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 18-65 year old of either gender

Exclusion Criteria:

* contraindication to regional block
* preexisting nerve damage
* hand or finger injury
* active skin infection
* allergy to local anesthetic
* disease states known to affect aquagenic skin wrinkling including cystic fibrosis, diabetic neuropathy, leprosy, vascular disease and diseases of autonomic function
* Patients with history of bleeding disorders or currently using anticoagulation agents
* contraindications to EMLA cream
* breaks in the skin on the finger EMLA is to be applied
* allergy to its constituents
* history of methemoglobinemia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2019-12-14 (Actual)

PRIMARY OUTCOMES:
Change in observed skin wrinkling | Assessed at baseline (prior to EMLA cream application) and 10, 20 and 30 minutes after its application
  Determined by judgements based on the "Wrinkling Assessment Scale" originally described by Ping Ng et. al. 2013: Grade 0: Wrinkling absent Grade 1: slight wrinkling and the fingertip is not smooth Grade 2: two or fewer lines of wrinkling on each side of the fingertip Grade 3: 3 or more lines of wrinkling on each side of the fingertip Grade 4: wrinkling completely distorts the pulp of the fingertip (see images presented in Wilder Smith et. al. 2015). A higher score indicates (3 or 4) full nerve function and the lower likelihood of nerve block. A lower score (0-2) indicate lower levels of nerve function and a higher likelihood of successful nerve blockade

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Collins, MD, Principal Investigator — Memorial University
Locations (1):
- Memorial University, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilder-Smith EP. Stimulated skin wrinkling as an indicator of limb sympathetic function. Clin Neurophysiol. 2015 Jan;126(1):10-6. doi: 10.1016/j.clinph.2014.08.007. Epub 2014 Sep 2. PMID 25216595
- [Background] Vasudevan TM, van Rij AM, Nukada H, Taylor PK. Skin wrinkling for the assessment of sympathetic function in the limbs. Aust N Z J Surg. 2000 Jan;70(1):57-9. doi: 10.1046/j.1440-1622.2000.01744.x. PMID 10696945